CLINICAL TRIAL: NCT02174926
Title: LASER Trial. LAparoscopic Elective Sigmoid Resection Following divERticulitis - a Multicenter, Prospective, Randomized Clinical Trial
Acronym: LASER
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Helsinki University Central Hospital (Other)
Responsible Party: Principal Investigator, Ville Sallinen, M.D., Ph.D., Helsinki University Central Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: LASERtrial
Record Dates: First submitted 2014-06-22; First posted 2014-06-26 (Estimated); Last update posted 2020-08-24 (Actual); Status verified 2020-08

CONDITIONS: Diverticulum; Colon, Sigmoid
MeSH Terms: conditions — Diverticulum | interventions — Conservative Treatment

ARMS (2):
- Conservative treatment (Active Comparator): Written lifestyle guidance and fiber supplements
  Interventions: Dietary Supplement: Conservative treatment
- Elective laparoscopic sigmoid resection (Experimental)
  Interventions: Procedure: Elective laparoscopic sigmoid resection

INTERVENTIONS:
Procedure: Elective laparoscopic sigmoid resection
  Arms: Elective laparoscopic sigmoid resection
Dietary Supplement: Conservative treatment — Written lifestyle guidance and fiber supplements
  Arms: Conservative treatment

SUMMARY:
The purpose of this study is to find out whether elective sigmoid resection will improve quality of life compared to conservative treatment with lifestyle guidance and fiber supplement in patients with a recurrent or complicated diverticulitis.

ELIGIBILITY:
Inclusion Criteria:

* Recurrent left colon diverticulitis (minimum 3 within 2 years, at least 1 confirmed with CT)

OR

* Earlier complicated left colon diverticulitis

OR

* Prolonged (over 3 months) pain or disturbance in bowel habits after a CT-confirmed left colon diverticulitis

Exclusion Criteria:

* Multimorbidity that prevents elective surgery
* Contraindication to laparoscopy
* Colonic stricture
* Fistula (e.g. colocutaneous, colovaginal, colovesical)
* Active malignancy
* Earlier resection of sigmoid colon or rectum
* Acute diverticulitis that has not settled
* Colonoscopy/sigmoidoscopy/virtual colonoscopy not performed within 2 years
* Age < 18 or > 75 years
* Pregnancy
* Inability to answer health surveys (e.g. dementia, psychiatric condition)

Ages: 18 Years to 75 Years | Sex: All
Age Groups: Adult, Older Adult
Enrollment: 133 (Estimated)
Dates: Start 2014-09 (Actual); Primary Completion 2019-04 (Actual); Study Completion 2027-12 (Estimated)

PRIMARY OUTCOMES:
Gastrointestinal quality of life-index change at 6 months | 6 months from randomization
  Difference in gastrointestinal quality of life-index (GIQLI) at randomization and 6 months from randomization.

SECONDARY OUTCOMES:
GIQLI at 12, 24, 48, and 96 months | 12, 24, 48, and 96 months from randomization
Short form (SF) 36 Health survey score at 6, 12, 24, 48, and 96 months | 6, 12, 24, 48, and 96 months from randomization
Recurrence and severity of recurrent diverticulitis | 0 - 96 months from randomization
Need of emergency surgery due to diverticulitis | 0 - 96 months from randomization
  Whether or not patient has undergone emergency surgery due to diverticulitis during follow-up period. Assessment will be carried out by patient questionnaire and search for patient records.
Need of elective sigmoid resection due to diverticulitis (conservative arm) | 0 - 96 months from randomization
  Whether or not patient has undergone elective sigmoid resection due to diverticulitis during follow-up period. Assessment will be carried out by patient questionnaire and search for patient records.
Complications due to elective sigmoid resection | 0 - 96 months from randomization
Mortality | 0 - 96 months
Complications of diverticular disease | 0 - 96 months
Stoma rate | 0 - 96 months from randomization

CONTACTS AND LOCATIONS:
Overall Officials: Ville Sallinen, M.D., Ph.D., Principal Investigator — Helsinki University Central Hospital
Locations (11):
- Finland (11):
  - Helsinki University Central Hospital, Jorvi Hospital, Espoo
  - Kanta-Häme Central Hospital, Hämeenlinna
  - Helsinki University Central Hospital, Helsinki
  - North Carelia Central Hospital, Joensuu
  - Keski-Suomi Central Hospital, Jyväskylä
  - Kuopio University Central Hospital, Kuopio
  - Päijät-Häme Central Hospital, Lahti
  - Oulu University Hospital, Oulu
  - Etelä-Pohjanmaa Central Hospital, Seinäjoki
  - Turku University Central Hospital, Turku
  - Vaasa Central Hospital, Vaasa

REFERENCES:
- [Derived] Santos A, Mentula P, Pinta T, Ismail S, Rautio T, Juusela R, Lahdesmaki A, Scheinin T, Sallinen V. Sigmoid Resection vs Conservative Treatment After Diverticulitis: Prespecified 4-Year Analysis of the LASER Randomized Clinical Trial. JAMA Surg. 2025 Jun 1;160(6):615-622. doi: 10.1001/jamasurg.2025.0572. PMID 40202724
- [Derived] Santos A, Mentula P, Pinta T, Ismail S, Rautio T, Juusela R, Lahdesmaki A, Scheinin T, Sallinen V. Quality-of-Life and Recurrence Outcomes Following Laparoscopic Elective Sigmoid Resection vs Conservative Treatment Following Diverticulitis: Prespecified 2-Year Analysis of the LASER Randomized Clinical Trial. JAMA Surg. 2023 Jun 1;158(6):593-601. doi: 10.1001/jamasurg.2023.0466. PMID 37074706
- [Derived] Santos A, Mentula P, Pinta T, Ismail S, Rautio T, Juusela R, Lahdesmaki A, Scheinin T, Sallinen V. Comparing Laparoscopic Elective Sigmoid Resection With Conservative Treatment in Improving Quality of Life of Patients With Diverticulitis: The Laparoscopic Elective Sigmoid Resection Following Diverticulitis (LASER) Randomized Clinical Trial. JAMA Surg. 2021 Feb 1;156(2):129-136. doi: 10.1001/jamasurg.2020.5151. PMID 33206182